CLINICAL TRIAL: NCT04025112
Title: Randomized Clinical Trial Comparing Rehabilitation Robotic Versus Conventional in Postoperative Period of Patients Submitted to Surgical Treatment of Breast Cancer
Brief Title: Randomized Clinical Trial Comparing Rehabilitation Robotic Versus Conventional After Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1563/2018
Record Dates: First submitted 2019-04-22; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Rehabilitation; Robotics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Armeo (Experimental): Patients group (54 patients) for robotic therapy.
  Interventions: Device: Armeo®Power
- Conventional (Active Comparator): Patients group (54 patients) for conventional rehabilitation protocol.
  Interventions: Other: Conventional rehabilitation protocol

INTERVENTIONS:
Device: Armeo®Power — Randomized patients will be offered rehabilitation robotic using Armeo®Power from Hocoma, the first robotic arm exoskeleton for integrated arm and hand therapy, during one month, three times a week, totalizing 12 sessions of 45 minutes.
  Arms: Armeo
Other: Conventional rehabilitation protocol — Randomized patients will be offered the conventional rehabilitation protocol from Barretos Cancer Hospital during one month, three times a week, totalizing 12 sessions of 45 minutes.
  Arms: Conventional

SUMMARY:
The aim of this study is to evaluate the effects of rehabilitation robotics in upper limb functionality involved in the surgical treatment of breast cancer. The study will be conducted following the delineation of randomized clinical trial. It will be assessed 108 women aged between 30 and 60 years, submitted to surgical treatment of breast cancer and axillary dissection.

DETAILED DESCRIPTION:
Breast cancer is one of the most common neoplasia types, with greater involvement in the female population, showing a high mortality rate in Brazil, due to diagnosis in advanced stages. With the increased survival of women treated for breast cancer, the evaluation of the effect of therapeutic resources for the morbidities resulting from surgical treatment of breast cancer are essential. The aim of this study is to evaluate the effects of rehabilitation robotics in upper limb functionality involved in the surgical treatment of breast cancer. The study will be conducted following the delineation of randomized clinical trial. It will be assessed 108 women aged between 30 and 60 years submitted to surgical treatment of breast cancer and axillary dissection, divided between two equal groups: control group (GC) - composed of women who had undergone conventional rehabilitation and experimental group (GE) - composed of women who had undergone rehabilitation robotics. The data obtained in the study aim to improve the forms of intervention against the functional alterations resulting from surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women submitted to quadrantectomy, simple mastectomy, radical mastectomy or modified radical mastectomy with complete axillary dissection.
* Women from 30 to 60 years old.
* Postoperatory range from 20 to 80 days.

Exclusion Criteria:

* Bilateral surgery
* Radiotherapy treatment in progress
* Upper limb metastasis

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast cancer in women
Enrollment: 108 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain classification change | "15 days" and "30 days"
  Pain measure will be done through Shoulder Pain and Disability Index (SPADI) questionnaire, classifying it from 0 (low) to 100 (high).
Arm strength change | "15 days" and "30 days"
  Arm strength measure will be performed with a hand dynamometer.
Change in the amplitude of arm movement | "15 days" and "30 days"
  The amplitude of arm movement wil be measured by a goniometer.
Upper limb disability change | "15 days" and "30 days"
  This outcome wil be measured by Disability of the Arm, Shoulder and Hand (DASH) questionnaire, classifying it from 0 (low) to 100 (high).

SECONDARY OUTCOMES:
Quality of life change | "15 days" and "30 days"
  Quality of life will be assessed by Functional Assessment of Cancer Therapy-Breast (FACT B+4) questionnaire.